CLINICAL TRIAL: NCT04015882
Title: Effects of Virtual Reality Exercises on Total Body Fat Ratio and Bone Health in Children With Acute Lymphoblastic Leukemia at Remitted
Brief Title: Effects of Exercises on Total Body Health in Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BezmialemVUb
Record Dates: First submitted 2018-07-13; First posted 2019-07-11 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia; Bone Density Increased
Keywords: acute lymphoblastic leukemia; bone density; total fat; exercise
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Osteosclerosis; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Active Comparator): the exercise group will applied virtual reality exercises by Nintendo Wii Fit Plus System Game Console.
  Interventions: Other: Exercise therapy
- control (No Intervention): No exercise applied the control group.

INTERVENTIONS:
Other: Exercise therapy — The exercise therapy group will make by physiotherapist supervision.
  Arms: exercise

SUMMARY:
In recent years, the survival of patients has increased with the success of leukemia treatment in children. However, according to the treatment modalities applied, complications such as changes in body composition such as obesity, osteoporosis and impaired bone health such as increased fragility are more frequent after treatment in patients.In this study, virtual reality exercise practices in remission of acute lymphoblastic leukemia cases will prevent negative effects on bone health and body composition and increase the quality of life of patients.

DETAILED DESCRIPTION:
Treatment and intervention options are being tried to avoid such complications that affect the quality of life of patients and there is still no standard treatment to convert bone health to healthy bone structure before the disease. There is a positive effect of improving the bone health of the activity and exercise programs. In this study, it was planned to demonstrate the positive effects of these changes on bone health through changes of adipokines and myokins released from fat and muscle tissue by virtual reality exercise method. Thus, the quality of life can be increased and cancer complications can be reduced in cancer cases.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for acute lymphoblastic leukemia
* At remitted term
* Being between 3 and 18 years
* Healthy cases of age and gender control group cases

Exclusion Criteria:

* Smaller than 3 years old and older than 18 years old
* Having a chronic illness
* Any drug use
* Any developmental anomaly

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
body mass index | 12 weeks
  Weight status among children and adolescents aged 2 through 19 years is defined based on BMI. In children and adolescents, overweight is defined as at or above the sex-specific 85th percentile on the CDC's 2000 BMI-for-age growth charts but less than the 95th percentile; obesity is defined as a BMI at or above the sex-specific 95th percentile.

SECONDARY OUTCOMES:
total body fat ratios | 12 weeks
  The methods have not been extensively studied in children. The method which provides the most useful measure of fat distribution remains to be determined. Dual-energy x-ray absorptiometry (DEXA) has been shown to be a reliable and accurate method of measuring fat mass
subcutaneous thickness | 12 weeks
  Anthropometric measures such as waist circumference provide simple means of estimating fat distribution that supplement measures of excess adiposity such as BMI, but ultimately cannot definitively differentiate between visceral and subcutaneous adipose tissue
bone mineral densities | 12 weeks
  Complications such as growth hormone deficiency and musculoskeletal deformity have negative effects on bone metabolism. Low bone mineral density is associated with fractures, skeletal deformity, pain, and substantial financial burden not only for childhood cancer survivors but also for public health care systems.
markers of bone metabolism | 12 weeks
  Normal pediatric reference ranges for serum markers of bone formation and resorption are a prerequisite for the assessment of metabolic bone disorders and for the monitoring of antiresorptive therapy or disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No